CLINICAL TRIAL: NCT03066323
Title: Effect of Tea Extract on Post Prandial Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: REF-BEV-2731
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Healthy
Keywords: Blood glucose
MeSH Terms: interventions — Tea

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tea extract (Active Comparator): Rice with tea extract
  Interventions: Other: Rice with tea extract
- No tea extract (Placebo Comparator): Rice without tea extract
  Interventions: Other: Rice without tea extract

INTERVENTIONS:
Other: Rice with tea extract — Rice with tea extract
  Arms: Tea extract
Other: Rice without tea extract — Rice without tea extract
  Arms: No tea extract

SUMMARY:
This study is designed as a randomized, single blind (data evaluation), placebo controlled, full cross-over study and conducted in 166 (including 10% drop out) males and females, aged ≥ 18 and ≤ 65 and waist circumference of >80 cm for women and >94 cm for men (indicating increased risk of metabolic complications (WHO)) and having a sedentary lifestyle. Subjects will receive rice with a tea extract and rice without a tea extract.

There will be three visits to the test facility: one screening visit and two intervention visits. During the intervention visits venous blood samples will be collected for the analysis of plasma glucose (t = -30m, -5m, 15m, 30m, 45m, 1h, 1h 30m, 2h and 3h, relative to the start of rice consumption ) and serum insulin (t = -5m, 30m, 1h, 2h and 3h).

Between the two intervention visits subjects have an interval of one week. This interval is required to minimize subject discomfort from repeated blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference > 80 cm for women and > 94 cm for men;
* Apparently healthy: no medical conditions which might affect the study measurements, absorption, metabolism and distribution (including diabetes type 1 and type 2, gastrointestinal dysfunction, gastrointestinal surgery and inflammatory diseases);
* Fasting blood glucose value of subjects is ≥ 3.4 and <6.1 mmol/litre (i.e. 62- 110 mg/dl) at screening;
* Being physically inactive (meaning less than five times 30 minutes of moderate activity per week, or less than three times 20 minutes of vigorous activity per week, or equivalent);

Exclusion Criteria:

* Use of antibiotics within 3 months before first intake of test product;
* Use of any other medication except paracetamol, within 14 days before first intake of test product;
* Consumption of > 14 units (female subjects) and > 21 units (male subjects) alcoholic drinks in a typical week;
* Dislike, known allergy or intolerance to the treatments or other food products provided during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Incremental area under the plasma glucose versus time curve | 0-2 hours

SECONDARY OUTCOMES:
Incremental area under the plasma glucose versus time curve | 0-3 hours
Maximum venous glucose concentration | 0-3 hours
Total area under the post prandial insulin versus time curves | 0-2 hours
Total area under the post prandial insulin versus time curves | 0-3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Fergus Shanahan, Prof, Principal Investigator — Consultant Gastroenterologist
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No